CLINICAL TRIAL: NCT01839266
Title: Prognostic Factors for Acute Pulmonary Embolism in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0034
Record Dates: First submitted 2013-04-01; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Acute Pulmonary Embolism (PE)
Keywords: acute PTE, prognostic factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute PE survivor, acute PE nonsurvivor: acute PE survivor, acute PE nonsurvivor (in-hospital death)

SUMMARY:
Acute pulmonary embolism (PE) is an important cause of in-hospital mortality and may be rapidly fatal if not diagnosed and treated. Despite recent advances in diagnostic and therapeutic modalities, it is still one of the important causes of hospital mortality. Previous several reports have described the variable outcome of patients with PE with reported mortality rate ranging from 8.1% (stable patients) to 25% (with cardiogenic shock) and 65% (post cardiopulmonary resuscitation). Nevertheless, there are no published studies from Korean hospitals that assessed the outcome of acute PE treated in the hospital with IV unfractionated heparin. We conducted this study to determine the outcome, risk factors, clinical characteristics and demographics of patients with acute PE and to identify possible demographic and clinical factors associated with prognosis.

ELIGIBILITY:
Inclusion Criteria:

patients admitted to the Severance Hospital, Yonsei University Health System with primary diagnosis of PE between January 2008 and December 2012. (diagnosed by CT and treated in the hospital with IV unfractionated heparin)

Exclusion Criteria:

1. diagnosis was prior to arrivalor
2. anticoagulation was contraindicated
3. diagnosis was not confirmed by CT

Min Age: 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute pulmonary embolism(PE) (diagnosed by CT) treated in the hospital with IV unfractionated heparin
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
prognostic factors of overall survival | change of acute pulmonary embolism(PE) for duration of hospital stay an expected average of 12 months
  In-hospital all-cause mortality with acute pulmonary embolism(PE) treated in the hospital with IV unfractionated heparin

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Chief of ICUs, Severance Hospital, Yonsei University Health System, Seoul, Seoul, South Korea